CLINICAL TRIAL: NCT04636450
Title: Comparison Between Manual and Rotatory Instrumentation Pulpectomy Treatments in Primary Mandibular Molars
Brief Title: Manual and Rotatory Instrumentation Pulpectomy in Primary Mandibular Molars
Acronym: RotaPulp
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Guanajuato (Other)
Collaborators: Universidad Latinoamericana (Unknown); University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Jaime Daniel Mondragón Uribe, Medical researcher, Universidad de Guanajuato
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ULA-2020-ODP-1
Record Dates: First submitted 2020-11-10; First posted 2020-11-19 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Dental Pulp Disease
Keywords: Pulp therapy; Rotatory system; Primary mandibular molar; Dental pulp cavity
MeSH Terms: conditions — Dental Pulp Diseases; Dental Caries

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Only the outcome assessor will be blinded as the interventions can not be blinded to the participant and care provider.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Adult manual instrumentation (Active Comparator): Primary mandibular molars who are treated with a manual pulpectomy and a K-file system.
  Interventions: Procedure: Manual pulpectomy
- Pediatric manual instrumentation (Experimental): Primary mandibular molars treated with a manual pulpectomy and a Kedo-SH system.
  Interventions: Procedure: Manual pulpectomy
- Adult rotatory instrumentation (Active Comparator): Primary mandibular molars treated with a rotatory technique pulpectomy and a K3 system.
  Interventions: Procedure: Rotatory technique pulpectomy
- Pediatric rotatory instrumentation (Experimental): Primary mandibular molars treated with a rotatory technique pulpectomy and a Kedo-S system
  Interventions: Procedure: Rotatory technique pulpectomy

INTERVENTIONS:
Procedure: Rotatory technique pulpectomy — Primary mandibular molars treated with a rotatory technique pulpectomy and a K3 system or a Kedo-S system.
  Arms: Adult rotatory instrumentation; Pediatric rotatory instrumentation
Procedure: Manual pulpectomy — Primary mandibular molars treated with a manual pulpectomy and a K-file system or a Kedo-SH system.
  Arms: Adult manual instrumentation; Pediatric manual instrumentation

SUMMARY:
In this study, the aim is to compare manual and rotatory pulpectomy techniques on 100 primary mandibular molars on children between the ages of 4 and 8 years. The plan is to conduct a randomized controlled trial with a 1:1 ratio for group allocation at a teaching university pediatric dentistry clinic between January 2021 and December 2021. Two manual systems, as well as two rotary systems, will be randomly assigned. The adult manual system used will be K-file and the adult rotary system will be K3. The pediatric manual system used in this study will be Kedo-SH, while the pediatric rotary system will be Kedo-S. The observed outcome measures in this study are the following: 1) instrumentation and filling time; 2) filling quality by radiographic evaluation; 3) postoperative pain levels using the visual analog scale at 12 and 24 hours; and 4) frequency of complications (e.g. fistulas, thinning of the mesiodistal walls, periapical or furcation radiolucency) after a 3-, 6-, 9-, and 12-month follow-up.

DETAILED DESCRIPTION:
Introduction

Dental caries is a prevalent chronic disease, affecting 60-90% of school-age children in industrialized countries; although in the last four decades the prevalence and severity of caries lesions have decreased, it is still a frequent disease for this age group. The American Dental Association (ADA) classifies dental caries by clinical presentation as initial, moderate, and severe; furthermore, the ADA classifies the disease using the international caries detection and diagnosis system (ICDAS II; International Caries Detection and Assessment System II) and by a radiographic presentation of the proximal faces based on the E0-E2, D1-D3 notation system. Within the non-vital pulp treatments, pulpectomy is indicated in temporary teeth; pulpectomy is a conventional endodontic treatment for teeth with exposed, infected, and/or necrotic tissue to eliminate pulp and periradicular infection.

In a recent systematic review that compared three different strategies for the management of deep caries lesions (i.e. complete caries removal, selective caries removal, and step caries removal), Aïem and colleagues (2020) report an increased restoration failure risk when selective removal is used compared to complete removal of caries. In a study where French dentists were surveyed on the management of deep caries lesions in primary dentition, the majority of respondents mentioned performing deep caries removal in a single step. Endodontic procedures in the pediatric population can assist to keep temporary teeth until exfoliation, which is a key principle of pediatric dentistry. Vital pulp and non-vital pulp treatments are employed in the treatment of severe lesions and deep caries; meanwhile, pulpectomy is a treatment largely used in the primary dentition. In pulp therapy, a pulpotomy is performed by removing the pulp from the chamber, while in a pulpectomy, all the tissue from both the chamber and the root canals is removed.

There are two parameters used to determine root canal treatment success: 1) the morphology and shaping of the canal; and 2) the duct cleanliness or the adequate level of disinfection provided by the type and quantity of intra-canal irrigation (e.g. chlorhexidine, sodium hypochlorite, citric acid, profuse irrigation). A pulpectomy is the technique of choice for primary dentition in deep carious lesions with pulp necrosis since pulpectomy has a higher success rate than pulpotomy. While the time for access to the root canal is less with the use of rotary instrumentation systems compared to a manual technique, manual techniques have the same efficacy as rotary systems in root canal cleaning procedures. Rotary systems have greater clinical success compared to manual techniques, in addition to having advantages in instrumentation time, canal shaping, reduction in working time, better cooperation and less patient fatigue, improvement in the conicity of the root canal, and promoting a higher quality of obturation. In a recent meta-analysis, Manchanda and colleagues (2020) conclude that rotary instrumentation has similar clinical and radiographic success rates to manual techniques in primary dentition; additionally, rotatory techniques show lower levels of postoperative pain and less instrumentation time. In the only study in the Mexican population that compared a rotary system (i.e. K3) against a manual technique (i.e. K-file) it was found that the instrumentation and obturation time was shorter, being a promising technique in children.

Given the limited comparative literature about rotatory techniques used in pulpectomy treatment, it is necessary to conduct clinical trials that compare both manual and rotatory techniques in first dentition treatment. So far, studies have been carried out comparing rotary systems designed for adults in the pediatric population. Recently, interest to validate and implement safe and effective protocols for the management of rotary systems in primary dentition has emerged in pediatric dentistry. Below is a protocol designed to investigate the advantages and disadvantages associated with the use of rotary systems designed for our population of interest.

Study design

Population: patients with pulpectomy indication according to the criteria mentioned by Kuo and colleagues (2006).

Place: Pediatric Dentistry Clinic, Universidad Latinoamericana, Campus Valle.

Time frame: January 2021 - December 2021

Sampling technique: convenience sampling with group randomization.

Study groups: 4 (n= 100 teeth)

1. Patients who are treated with a manual pulpectomy and a K-file system.
2. Patients who are treated with a manual pulpectomy and a Kedo-SH system.
3. Patients who are treated with a rotatory technique pulpectomy and a K3 system.
4. Patients who are treated with a rotatory technique pulpectomy and a Kedo-S system.

PICOS framework

P: pediatric population

I: manual system pulpectomy

C: rotary system pulpectomy

O: instrumentation and obturation time, filling quality by radiographic evaluation, postoperative pain levels at 12hr and 24hr, frequency of complications (e.g. fistulas, thinning of the mesiodistal walls, periapical or furcation radiolucency) after a 3-, 6-, 9-, and 12-month follow-up.

S: a randomized controlled trial

Research question

Are there differences between the use of a manual system compared to a rotary system in the pediatric population?

Main objective

Compare the performance between a manual technique and a rotatory technique during biomechanical work.

Particular objectives

1. Compare the instrumentation (i.e. during biomechanical work) and filling time between a manual technique and a rotatory technique.
2. Compare the filling quality by radiographic evaluation between a manual technique and a rotatory technique at the end of the procedure.
3. Compare postoperative pain levels using the visual analog scale at 12 and 24 hours.
4. Compare the frequency of complications (e.g. fistulas, thinning of the mesiodistal walls, periapical or furcation radiolucency) after a 3-, 6-, 9-, and 12-month follow-up between the two techniques.

Hypotheses

H1: The rotatory techniques will take less instrumentation and obturation time than the manual techniques.

H1: The quality of the obturation in the rotatory technique will be reported radiographically more frequently as optimal than the manual technique.

H1: The pain levels reported by patients will be lower in the rotatory technique than in the manual technique.

H1: The rotatory technique will have a lower frequency of complications such as fistulas, thinning of the mesiodistal walls, periapical or furcation radiolucency at each time point compared to the manual technique.

Statistical analysis

Descriptive statistics will be performed on all variables. Statistical analysis will be performed using SPSS 25 (SPSS Inc., Chicago, IL). All variables will be examined to determine the existence of outliers and whether or not they meet the Gaussian distribution assumption; furthermore, Gaussian distribution will be determined with the Shapiro-Wilk test and by visualizing the data through histograms and Q-Q graphs. The demographic and clinical variables will be summarized in proportions and percentages. Nominal variables will be evaluated with Chi-square tests to assess differences between groups. Categorical variables will be evaluated to determine statistical inferences with the Mann-Whitney test. Continuous variables will be assessed for statistical inferences using t-tests and Levene's test to assess variance equality. Statistical significance will be set at p= 0.05 and a Bonferroni correction will be made for multiple comparisons.

Sample size

The sample size necessary to detect statistically significant differences was calculated by taking the following parameters; α = 0.05 and statistical power of 0.8 (i.e. 1-β). For the calculation of the sample size, the time of instrumentation was used as a measure of clinical outcome. The sample was calculated based on the article by Ochoa-Romero and colleagues (2011) where instrumentation time was used as the primary outcome. The sample calculator used can be found on the website: https://clincalc.com/stats/samplesize.aspx. The calculator designed for two independent groups for continuous variables was selected, using the mean for each group (i.e. group 1: rotatory technique 1.7 minutes ± 0.5; group 2: manual technique 2.5 minutes ± 0.8) taking into account an enrollment 1:1 ratio for this study. The total sample size was 24 teeth (i.e. at least 6 teeth per group to find statistically significant differences in instrumentation time).

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 4 to 8 years old.
2. Both genders.
3. Patients with an indication for pulpectomy for mandibular molars, based on the of Kuo and colleagues criteria (2006).
4. Patients requiring pulpectomy in posterior teeth.
5. Adequate dental structure of the crown.
6. Patients with a remnant structure of at least two-thirds of the root.
7. Patients with a medical file at the Pediatric Dentistry Clinic, Universidad Latinoamericana, Campus Valle.
8. Patients with signed informed consent.

Exclusion Criteria:

1. Patients requiring pulpotomy, extraction, or pulp regeneration therapy.
2. Patients who are older than 9 years.
3. An unrestorable tooth.
4. Internal resorption in the roots visible on radiographs.
5. Teeth with mechanical or carious perforations of the floor of the pulp chamber.
6. Excessive pathologic root resorption involving more than a third of the root.
7. Excessive pathologic loss of bone support, with loss of the normal periodontal attachment.
8. Presence of a dentigerous or follicular cyst.
9. Periapical or interradicular lesion involving the crypt of the developing permanent successor.
10. Patients with the diagnosis of molar incisor hypomineralization (MIH).
11. Patient's whose legal guardian does not provide their informed consent to participate in this study.
12. Uncooperative patients.

Elimination criteria

a. Patients who do not complete the treatment or radiographic follow-up at least at a cut-off point.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2020-12-08 (Actual); Primary Completion 2021-12-15 (Estimated); Study Completion 2022-07-15 (Estimated)

PRIMARY OUTCOMES:
Instrumentation time | Minutes; intraoperative time.
  The time needed to shape the root canal.
Obturation time | Minutes, intraoperative time.
  Time needed to obturate the root canals.
Filling quality | Immediately after surgical procedure.
  Radiographic evaluation of the root canal filling.
Postoperative pain | 12 hours
  Pain resulting from the surgical procedure, evaluated with the visual analog pain scale (range, 1 to 10; the higher the score the worst the outcome).
Postoperative pain | 24 hours
  Pain resulting from the surgical procedure, evaluated with the visual analog pain scale (range, 1 to 10; the higher the score the worst the outcome).

SECONDARY OUTCOMES:
Complications secondary to procedure | 3-months
  Frequency of fistulas, thinning of the mesiodistal walls, periapical or furcation radiolucency, among other possible complications
Complications secondary to procedure | 6-months
  Frequency of fistulas, thinning of the mesiodistal walls, periapical or furcation radiolucency, among other possible complications
Complications secondary to procedure | 9-months
  Frequency of fistulas, thinning of the mesiodistal walls, periapical or furcation radiolucency, among other possible complications
Complications secondary to procedure | 12-months
  Frequency of fistulas, thinning of the mesiodistal walls, periapical or furcation radiolucency, among other possible complications

CONTACTS AND LOCATIONS:
Overall Officials: Benjamín Franco Sánchez, DDS, Principal Investigator — Universidad Latinoamericana; Marianela Hernández-Baños, DDS, Principal Investigator — Universidad Latinoamericana; Jaime D Mondragon, MD, MSc, Principal Investigator — University Medical Center Groningen, Universidad de Guanajuato
Locations (1):
- Clínica de Odontopediatría, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
All anonymized patient data will be made available upon request.
Supporting Information: Study Protocol, SAP
Time Frame: At the conclusion of the study.
Access Criteria: Access granted by the principal investigators.

REFERENCES:
- [Result] Aiem E, Joseph C, Garcia A, Smail-Faugeron V, Muller-Bolla M. Caries removal strategies for deep carious lesions in primary teeth: Systematic review. Int J Paediatr Dent. 2020 Jul;30(4):392-404. doi: 10.1111/ipd.12616. Epub 2020 Feb 18. PMID 31943437
- [Result] Anusavice KJ. Present and future approaches for the control of caries. J Dent Educ. 2005 May;69(5):538-54. PMID 15897335
- [Result] Casas MJ, Kenny DJ, Johnston DH, Judd PL. Long-term outcomes of primary molar ferric sulfate pulpotomy and root canal therapy. Pediatr Dent. 2004 Jan-Feb;26(1):44-8. PMID 15080357
- [Result] Crespo S, Cortes O, Garcia C, Perez L. Comparison between rotary and manual instrumentation in primary teeth. J Clin Pediatr Dent. 2008 Summer;32(4):295-8. doi: 10.17796/jcpd.32.4.l57l36355u606576. PMID 18767460
- [Result] Frencken JE, Sharma P, Stenhouse L, Green D, Laverty D, Dietrich T. Global epidemiology of dental caries and severe periodontitis - a comprehensive review. J Clin Periodontol. 2017 Mar;44 Suppl 18:S94-S105. doi: 10.1111/jcpe.12677. PMID 28266116
- [Result] Fuks AB. Pulp therapy for the primary and young permanent dentitions. Dent Clin North Am. 2000 Jul;44(3):571-96, vii. PMID 10925773
- [Result] Fuks, A.B., Guelmann, M., Kupietzky, A. (2012). Current developments in pulp therapy for primary teeth. Endodontic Topics, 23, 50-72. https://doi.org/10.1111/etp.12003
- [Result] Hecksher F, Vidigal B, Coelho P, Otoni D, Alvarenga C, Nunes E. Endodontic Treatment in Artificial Deciduous Teeth through Manual and Mechanical Instrumentation: A Pilot Study. Int J Clin Pediatr Dent. 2019 Jan-Feb;12(1):15-17. doi: 10.5005/jp-journals-10005-1581. PMID 31496565
- [Result] Kaur, R., Singh, R., Sethi, K., Garg, S., Miglani, S. (2014). Review article irrigating solutions in Pediatric Dentistry: literature review and update. J Adv Med Dent Sci, 2, 104- 115.
- [Result] Kher, M.S., Rao, A. Pulp therapy in primary teeth. Clin Dent Rev 4, 16 (2020). https://doi.org/10.1007/s41894-020-00081-z
- [Result] Lopes-Fatturi, Aluhê, Souza, Juliana Feltrin de, Menezes, José Vitor Nogara Borges, Fraiz, Fabian Calixto, & Assunção, Luciana Reichert da Silva. (2020). A Survival Analysis of Different Pulp Therapies in Decayed Primary Teeth. Pesquisa Brasileira em Odontopediatria e Clínica Integrada, 20, e4822. Epub April 27, 2020. https://dx.doi.org/10.1590/pboci.2020.038
- [Result] Manchanda S, Sardana D, Yiu CKY. A systematic review and meta-analysis of randomized clinical trials comparing rotary canal instrumentation techniques with manual instrumentation techniques in primary teeth. Int Endod J. 2020 Mar;53(3):333-353. doi: 10.1111/iej.13233. Epub 2019 Nov 26. PMID 31587323
- [Result] Muller-Bolla M, Garcia A, Aiem E, Domejean S. Dentists' decisions for deep carious lesions management in primary teeth. Int J Paediatr Dent. 2020 Sep;30(5):578-586. doi: 10.1111/ipd.12639. Epub 2020 Apr 7. PMID 32189409
- [Result] Ochoa-Romero T, Mendez-Gonzalez V, Flores-Reyes H, Pozos-Guillen AJ. Comparison between rotary and manual techniques on duration of instrumentation and obturation times in primary teeth. J Clin Pediatr Dent. 2011 Summer;35(4):359-63. doi: 10.17796/jcpd.35.4.8k013k21t39245n8. PMID 22046692
- [Result] Panchal V, Jeevanandan G, Erulappan SM. Comparison between the Effectiveness of Rotary and Manual Instrumentation in Primary Teeth: A Systematic Review. Int J Clin Pediatr Dent. 2019 Jul-Aug;12(4):340-346. doi: 10.5005/jp-journals-10005-1637. PMID 31866721
- [Result] Petersen PE, Bourgeois D, Ogawa H, Estupinan-Day S, Ndiaye C. The global burden of oral diseases and risks to oral health. Bull World Health Organ. 2005 Sep;83(9):661-9. Epub 2005 Sep 30. PMID 16211157
- [Result] Pozos-Guillen A, Garcia-Flores A, Esparza-Villalpando V, Garrocho-Rangel A. Intracanal irrigants for pulpectomy in primary teeth: a systematic review and meta-analysis. Int J Paediatr Dent. 2016 Nov;26(6):412-425. doi: 10.1111/ipd.12228. Epub 2016 Feb 22. PMID 26898157
- [Result] Rawson TH, Rayes S, Strizich G, Salazar CR. Longitudinal Study Comparing Pulpectomy and Pulpotomy Treatments for Primary Molars of Alaska Native Children. Pediatr Dent. 2019 May 15;41(3):214-220. PMID 31171074
- [Result] Taylor GD, Vernazza CR, Abdulmohsen B. Success of endodontic management of compromised first permanent molars in children: A systematic review. Int J Paediatr Dent. 2020 May;30(3):370-380. doi: 10.1111/ipd.12599. Epub 2019 Dec 13. PMID 31778237
- [Result] Pulp Therapy for Primary and Immature Permanent Teeth. Pediatr Dent. 2017 Sep 15;39(6):325-333. No abstract available. PMID 29179372
- [Result] Young DA, Novy BB, Zeller GG, Hale R, Hart TC, Truelove EL; American Dental Association Council on Scientific Affairs; American Dental Association Council on Scientific Affairs. The American Dental Association Caries Classification System for clinical practice: a report of the American Dental Association Council on Scientific Affairs. J Am Dent Assoc. 2015 Feb;146(2):79-86. doi: 10.1016/j.adaj.2014.11.018. PMID 25637205